CLINICAL TRIAL: NCT06207331
Title: Effects of Atomized Dexmedetomidine on Lung Function in Patients With Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no patient enrolled.
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Bing Chen, Ph.D, Associate professor, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023.134
Record Dates: First submitted 2023-11-21; First posted 2024-01-17 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Function Tests; Chronic Obstructive Pulmonary Disease; Dexmedetomidine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Dexmedetomidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine 0.5 μg/kg (Experimental): Participants inhale 0.5 μg/kg dexmedetomidine prepared in 2 ml 0.9% saline.
- Dexmedetomidine 1 μg/kg (Experimental): Participants inhale 1 μg/kg dexmedetomidine prepared in 2 ml 0.9% saline.
- Placebo (Placebo Comparator): Participants inhale 2 ml atomized 0.9% saline.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine 0.5 μg/kg — Participants inhale the atomized 0.5 μg/kg dexmedetomidine in 2 ml of 0.9% saline.
  Other Names: Dexmedetomidine Hydrochloride
Drug: Dexmedetomidine 1 μg/kg — Participants inhale the atomized 1 μg/kg dexmedetomidine in 2 ml of 0.9% saline.
  Other Names: Dexmedetomidine Hydrochloride
Drug: Saline — Participants inhale atomized 2 ml 0.9% saline.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Studies have shown that intravenous infusion and nebulized dexmedetomidine can improve lung function in mechanically ventilated patients, including those with preoperative COPD, exerting lung protection. However, these studies are based on mechanical ventilation patients under general anesthesia, and more intuitive research is needed on whether dexmedetomidine can also exercise pulmonary precaution in awake patients. Pulmonary function monitoring is the most direct way to evaluate changes in lung function in awake patients. Portable pulmonary function machines can assess lung function in a variety of settings. In addition, compared with intravenous administration, nebulized inhalation administration directly acts on the mucosa of the respiratory tract, does not involve invasive operations, and has higher safety and comfort. Therefore, this study intends to use portable pulmonary function instruments and non-invasive ambulatory respiratory monitors to evaluate the effect of nebulized dexmedetomidine on lung function in COPD patients to guide the perioperative management of COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common respiratory disease that seriously endangers the physical and mental health of patients. Surgical patients with COPD will increase the risk of postoperative pulmonary complications and the risk of complications of extrapulmonary organs such as heart and kidney, and lead to prolonged hospital stay, increased medical costs, and increased perioperative mortality. Therefore, it is necessary to explore drugs with lung protection effects to improve the perioperative safety of COPD patients.

Dexmedetomidine (Dex) is a new type of highly selective α2-adrenergic receptor agonist, which has the effects of sedative-hypnotic, anti-inflammatory, stress reduction, hemodynamic stabilization, analgesia, and organ protection, and has little inhibitory effect on respiratory function. In recent years, studies have found that dexmedetomidine may have the effect of improving lung function. In addition, human studies have found that intravenous infusion of dexmedetomidine (loading dose 0.5 to 1 μg/kg or 0.5 to 0.7 μg/kg/hour) can reduce inflammation levels, improve oxidative stress, reduce plateau pressure, peak airway pressure, airway resistance, and improve lung compliance, thereby improving oxygenation and postoperative pulmonary complications, and promoting patient recovery. In obese patients undergoing laparoscopic gastric reduction, intraoperative intravenous dexmedetomidine infusion (loading dose of 1 μg/kg, followed by 1 μg/kg/hour) improves lung compliance and oxygenation. One study found that intraoperative intravenous infusion of dexmedetomidine (loading dose of 1 μg/kg, followed by 0.5 μg/kg/hour) increased forced expiratory volume in one second and improved postoperative oxygenation on days 1 and 2 after one-lung ventilation. Another study found that nebulized inhalation of 0.5 μg/kg, 1 μg/kg, and 2 μg/kg dexmedetomidine in one-lung ventilation for thoracic surgery improved lung compliance and oxygenation.

These studies have shown that intravenous infusion and nebulized dexmedetomidine can improve lung function in mechanically ventilated patients, including those with preoperative COPD, exerting lung protection. However, these studies are based on mechanical ventilation patients under general anesthesia, and more intuitive research is needed on whether dexmedetomidine can also exercise pulmonary precaution in awake patients. Pulmonary function monitoring is the most direct way to evaluate changes in lung function in awake patients. Portable pulmonary function machines can assess lung function in a variety of settings. In addition, compared with intravenous administration, nebulized inhalation administration directly acts on the mucosa of the respiratory tract, does not involve invasive operations, has limited effect, high safety, fewer side effects, and higher comfort. Therefore, this study intends to use portable pulmonary function instruments and non-invasive ambulatory respiratory monitors to evaluate the effect of nebulized dexmedetomidine on lung function in COPD patients to guide the perioperative management of COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosed COPD who are scheduled to undergo elective surgery (FEV1/FVC ratio< 0.70)
2. Patients with mild, moderate, and severe COPD (FEV1≥30% predicted)
3. Age ≥ 40 years old, ≤ 80 years old
4. American Society of Anesthesiologists (ASA) Physical Situation Grading I-III
5. Able to cooperate with the experiment, voluntarily participate and be able to understand and sign the informed consent form

Exclusion Criteria:

1. Obese patients (BMI>28 kg/m2)
2. Patients with grade 3 hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg)
3. Patients with myocardial infarction and shock in the past 3 months
4. Patients with unstable angina pectoris with NYHA heart function grade III or IV in the last 4 weeks
5. Tachycardia (heart rate >120 beats/min), bradycardia (heart rate <45 beats/min), and degree II or III atrioventricular block
6. Patients with severe or uncontrolled bronchial asthma, pulmonary infection, bronchiectasis, thoracic malformation, pneumothorax, hemothorax, giant pulmonary bulla, and massive hemoptysis in the last 4 weeks
7. Pulmonary artery pressure ≥60 mmHg
8. Patients with Child B or C liver function
9. Patients with stage 4 or 5 chronic kidney disease
10. Patients with hyperthyroidism and pheochromocytoma
11. Patients with seizures requiring medication
12. Pregnant women
13. Patients with tympanic membrane perforation
14. Patients allergic to dexmedetomidine;
15. For any reason, it is not possible to cooperate with the study or the researcher considers it inappropriate to be included in this experiment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
FVC | 10 minutes and 30 minutes after administration of nebulized drugs
  Forced vital capacity

SECONDARY OUTCOMES:
FEV1 | 10 minutes and 30 minutes after administration of nebulized drugs
  Forced expiratory volume in one second
FEV1/FVC% | 10 minutes and 30 minutes after administration of nebulized drugs
  Forced expiratory volume in one second/Forced vital capacity
MMEF | 10 minutes and 30 minutes after administration of nebulized drugs
  maximal mid-expiratory flow curve
PEF | 10 minutes and 30 minutes after administration of nebulized drugs
  Peak expiratory flow
BEV | 10 minutes and 30 minutes after administration of nebulized drugs
  Back-extrapolation volume
FET | 10 minutes and 30 minutes after administration of nebulized drugs
  Forced expiratory time
VC | 10 minutes and 30 minutes after administration of nebulized drugs
  Vital capacity
FEV1/VC | 10 minutes and 30 minutes after administration of nebulized drugs
  Forced expiratory volume in one second/vital capacity
FEF25%，FEF50%，FEF75%， | 10 minutes and 30 minutes after administration of nebulized drugs
  forced expiratory flow at 25%, 50%, and 75% of FVC exhaled
PIF | 10 minutes and 30 minutes after administration of nebulized drugs
  peak inspiratory flow
FIVC | 10 minutes and 30 minutes after administration of nebulized drugs
  forced inspiratory vital capacity
FIF25, FIF50, FIF75 | 10 minutes and 30 minutes after administration of nebulized drugs
  forced inspiratory flow at 25%, 50%, and 75% of FIVC
FIV1 | 10 minutes and 30 minutes after administration of nebulized drugs
  forced inspiratory volume in 1 second
MVV | 10 minutes and 30 minutes after administration of nebulized drugs
  maximal ventilatory volume
Richmond Agitation-Sedation Scale (RASS) | 10 minutes and 30 minutes after administration of nebulized drugs
  RASS is a 10-point scale, with four levels of anxiety or agitation (+1 to +4 [combative]), one level to denote a calm and alert state (0), and 5 levels of sedation (-1 to -5) culminating in unarousable (-5).
heart rate | 10 minutes and 30 minutes after administration of nebulized drugs
  heart rate (beat per min)
Systolic and diastolic blood pressures | 10 minutes and 30 minutes after administration of nebulized drugs
  Systolic and diastolic blood pressures (mmHg)
SPO2 | 10 minutes and 30 minutes after administration of nebulized drugs
  Pulse oximetry (SpO2)

CONTACTS AND LOCATIONS:
Overall Officials: Bing Chen, PhD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available with the corresponding author when required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available when we publish and keep it for five years.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Groeben H, Mitzner W, Brown RH. Effects of the alpha2-adrenoceptor agonist dexmedetomidine on bronchoconstriction in dogs. Anesthesiology. 2004 Feb;100(2):359-63. doi: 10.1097/00000542-200402000-00026. PMID 14739811
- [Background] Yamakage M, Iwasaki S, Satoh JI, Namiki A. Inhibitory effects of the alpha-2 adrenergic agonists clonidine and dexmedetomidine on enhanced airway tone in ovalbumin-sensitized guinea pigs. Eur J Anaesthesiol. 2008 Jan;25(1):67-71. doi: 10.1017/S0265021507002591. Epub 2007 Sep 21. PMID 17888193
- [Background] Di Bella C, Skouropoulou D, Stabile M, Muresan C, Grasso S, Lacitignola L, Valentini L, Crovace A, Staffieri F. Respiratory and hemodynamic effects of 2 protocols of low-dose infusion of dexmedetomidine in dogs under isoflurane anesthesia. Can J Vet Res. 2020 Apr;84(2):96-107. PMID 32255904
- [Background] Jiang H, Kang Y, Ge C, Zhang Z, Xie Y. One-lung ventilation patients: Clinical context of administration of different doses of dexmedetomidine. J Med Biochem. 2022 Apr 8;41(2):230-237. doi: 10.5937/jomb0-33870. PMID 35510198
- [Background] Kostroglou A, Kapetanakis EI, Matsota P, Tomos P, Kostopanagiotou K, Tomos I, Siristatidis C, Papapanou M, Sidiropoulou T. Monitored Anesthesia Care with Dexmedetomidine Supplemented by Midazolam/Fentanyl versus Midazolam/Fentanyl Alone in Patients Undergoing Pleuroscopy: Effect on Oxygenation and Respiratory Function. J Clin Med. 2021 Aug 9;10(16):3510. doi: 10.3390/jcm10163510. PMID 34441805
- [Background] Xia R, Xu J, Yin H, Wu H, Xia Z, Zhou D, Xia ZY, Zhang L, Li H, Xiao X. Intravenous Infusion of Dexmedetomidine Combined Isoflurane Inhalation Reduces Oxidative Stress and Potentiates Hypoxia Pulmonary Vasoconstriction during One-Lung Ventilation in Patients. Mediators Inflamm. 2015;2015:238041. doi: 10.1155/2015/238041. Epub 2015 Jul 26. PMID 26273134
- [Background] Hasanin A, Taha K, Abdelhamid B, Abougabal A, Elsayad M, Refaie A, Amin S, Wahba S, Omar H, Kamel MM, Abdelwahab Y, Amin SM. Evaluation of the effects of dexmedetomidine infusion on oxygenation and lung mechanics in morbidly obese patients with restrictive lung disease. BMC Anesthesiol. 2018 Aug 14;18(1):104. doi: 10.1186/s12871-018-0572-y. PMID 30103679
- [Background] Jannu V, Dhorigol MG. Effect of Intraoperative Dexmedetomidine on Postoperative Pain and Pulmonary Function Following Video-assisted Thoracoscopic Surgery. Anesth Essays Res. 2020 Jan-Mar;14(1):68-71. doi: 10.4103/aer.AER_9_20. Epub 2020 Mar 16. PMID 32843795
- [Background] Lee SH, Kim N, Lee CY, Ban MG, Oh YJ. Effects of dexmedetomidine on oxygenation and lung mechanics in patients with moderate chronic obstructive pulmonary disease undergoing lung cancer surgery: A randomised double-blinded trial. Eur J Anaesthesiol. 2016 Apr;33(4):275-82. doi: 10.1097/EJA.0000000000000405. PMID 26716866
- [Background] Xu B, Gao H, Li D, Hu C, Yang J. Nebulized dexmedetomidine improves pulmonary shunt and lung mechanics during one-lung ventilation: a randomized clinical controlled trial. PeerJ. 2020 Jun 5;8:e9247. doi: 10.7717/peerj.9247. eCollection 2020. PMID 32547872
- [Background] Yang L, Cai Y, Dan L, Huang H, Chen B. Effects of dexmedetomidine on pulmonary function in patients receiving one-lung ventilation: a meta-analysis of randomized controlled trial. Korean J Anesthesiol. 2023 Dec;76(6):586-596. doi: 10.4097/kja.22787. Epub 2023 Mar 16. PMID 36924790